CLINICAL TRIAL: NCT05928351
Title: Investigation of the Efficacy of Neuroscience Pain Education in Patients With Total Knee Arthroplasty
Brief Title: Pain Neuroscience Education in Patients With Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Abdulhamit Tayfur, Principal Investigator, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023/605
Record Dates: First submitted 2023-06-15; First posted 2023-07-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis, Knee
Keywords: pain neuroscience education; knee; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: the blinded assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNE Group (Experimental): Pain Neuroscience Education + Standard Physiotherapy Program
  Interventions: Other: Pain Neuroscience Education; Other: Standard Physiotherapy Program (SPP)
- Control Group (Active Comparator): Standard Physiotherapy Program
  Interventions: Other: Standard Physiotherapy Program (SPP)

INTERVENTIONS:
Other: Pain Neuroscience Education — The experimental group will follow a PNE protocol based on previous procedure for 6 weeks in addition to the standard physiotherapy program (SPP) in postoperative period.
  Each PNE session will take 45-60 min. PNE will be conducted in line with international guidelines and covered the neurophysiology of pain, transition from acute to chronic pain, and the nervous system ability to modulate the pain experience.
  Arms: PNE Group
Other: Standard Physiotherapy Program (SPP) — The control group will follow a SPP. The 45-minute-long treatment sessions will be held 5 days per week. The treatment program will be organized in 3 periods as 0-2 weeks, 3-4 weeks and 5-6 weeks. The overall treatment program will include scar massage, patellar mobilization, coldpack, ankle pump, quadriceps and hamstring strengthening, hip range of motion, hip strengthening exercises, squat, ascending and descending stairs, walking training. All exercises will be 10 repetitions x 2 sets.

SUMMARY:
The aim of Pain Neuroscience Education (PNE) is to explain to patients the biological and physiological processes involved in a pain experience and, more importantly, defocus the issues associated with the anatomical structures. PNE provides compelling evidence in reducing pain, disability, pain catastrophization, and limited physical movement in musculoskeletal problems. Knee osteoarthritis (KOA) is a very common painful musculoskeletal problem, especially in people over 50 years old, and lead to decrease in knee range of motion. Despite costly arthroscopic surgeries and long-term physiotherapy treatments, poor outcomes are common. The lack of satisfactory results suggests that some practices should be revised. Although PNE could be useful as an intervention, to our knowledge, there is no randomized controlled trial in the literature investigating the effects of PNE in patients with a KOA. Therefore, we aimed to examine the effectiveness of PNE on clinical outcomes in patients with KOA.

ELIGIBILITY:
Inclusion Criteria:

* Having a body mass index between 19-40 kg/m2,
* Having had a unilateral TKA,
* Knee pain score to be 4 and above daily according to the visual analog scale,
* Ability to read, speak and understand Turkish.

Exclusion Criteria:

* Prosthesis disorders requiring re-surgery,
* Having visual, auditory and cognitive impairment,
* Secondary TKA such as rheumatoid arthritis,
* Acute pain,
* Pregnancy, drug and alcohol use,
* Having bilateral TKA,
* Not volunteering to participate in the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pain severity | Baseline
  Visual Analogue Scale (0-10, higher means worse)
Pain severity change is being assessed | 6 week
  Visual Analogue Scale (0-10, higher means worse)
Pain and Function | Baseline
  Knee Injury and Osteoarthritis Outcome Score (0-100, higher means better)
Pain and Function change are being assessed | 6 week
  Knee Injury and Osteoarthritis Outcome Score (0-100, higher means better)
Pain and Function | Baseline
  Western Ontario and McMaster Universities Arthritis Index (0-96, higher means worse)
Pain and Function change are being assessed | 6 week
  Western Ontario and McMaster Universities Arthritis Index (0-96, higher means worse)

SECONDARY OUTCOMES:
Pain Catastrophizing | Baseline
  Pain Catastrophizing Scale (0-52, higher means worse)
Pain Catastrophizing change is being assessed | 6 week
  Pain Catastrophizing Scale (0-52, higher means worse)
Kinesiophobia | Baseline
  Tampa Scale of Kinesiophobia (17-68, higher means worse)
Kinesiophobia change is being assessed | 6 week
  Tampa Scale of Kinesiophobia (17-68, higher means worse)
Level of quality of life | Baseline
  Short Form-12 (0-100, higher means better)
Level of quality of life change is being assessed | 6 week
  Short Form-12 (0-100, higher means better)
Anxiety and Depression | Baseline
  Hospital Anxiety Depression Scale (0-21, higher means worse)
Anxiety and Depression change is being assessed | 6 week
  Hospital Anxiety Depression Scale (0-21, higher means worse)
Physical Function | Baseline
  40 meter walking test (in seconds, less is better)
Physical Function change is being assessed | 6 week
  40 meter walking test (in seconds, less is better)

CONTACTS AND LOCATIONS:
Locations (1):
- Ahi Evran University, Kırşehir, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Louw A PT, PhD, Zimney K PT, DPT, Reed J PT, DPT, Landers M PT, DPT, PhD, Puentedura EJ PT, DPT, PhD. Immediate preoperative outcomes of pain neuroscience education for patients undergoing total knee arthroplasty: A case series. Physiother Theory Pract. 2019 Jun;35(6):543-553. doi: 10.1080/09593985.2018.1455120. Epub 2018 Mar 28. PMID 29589782
- [Derived] Tayfur A, Ozyurt F, Kodak MI, Cakmak MF, Ozsoy G, Cigdem Karacay B, Ozsoy I, Basat HC, Kararti C. The efficacy of pain neuroscience education in patients after total knee arthroplasty: a single blind randomized controlled trial. Physiother Theory Pract. 2025 Dec;41(12):2513-2523. doi: 10.1080/09593985.2025.2526025. Epub 2025 Jul 1. PMID 40590360